CLINICAL TRIAL: NCT04199910
Title: 4beta-hydroksikolesteroli Maksakirroosissa
Brief Title: 4beta-hydroxycholesterol in Cirrhosis
Status: Suspended | Type: Observational
Why Stopped: COVID pandemia hinders recruitment
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Janne Hukkanen, Professor, University of Oulu
Other Study IDs: 4bHC kirroosissa
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Liver cirrhosis with spironolactone
  Interventions: Other: There is no intervention, only research blood samples are collected
- Liver cirrhosis with rifaximin
  Interventions: Other: There is no intervention, only research blood samples are collected
- Liver cirrhosis without spironolactone or rifaximin
  Interventions: Other: There is no intervention, only research blood samples are collected
- Pneumonia
  Interventions: Other: There is no intervention, only research blood samples are collected
- Crohn's disease
  Interventions: Other: There is no intervention, only research blood samples are collected
- Ulcerative colitis
  Interventions: Other: There is no intervention, only research blood samples are collected

INTERVENTIONS:
Other: There is no intervention, only research blood samples are collected — Research blood samples collected

SUMMARY:
The aim is to evaluate the levels of oxysterols and especially 4beta-hydroxycholesterol in patients with liver cirrhosis. Three cirrhosis cohorts are recruited: patients treated with spironolactone, patients treated with rifaximin, patients without spironolactone or rifaximin. Also three other control cohorts are recruited: patients with pneumonia, patients with Crohn's disease, patients with ulcerative colitis. The effect of the cirrhosis and its medications spironolactone and rifaximin are compared to control groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis, pneumonia, Crohn's disease or colitis ulcerosa
* Treated in the ward 42 of the Oulu University Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis, pneumonia, Crohn's disease or colitis ulcerosa treated in the ward 42 of the Oulu University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood 4beta-hydroxycholesterol concentration | At the time point of the blood collection - cross-sectional. One day.
  Blood 4beta-hydroxycholesterol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Undecided